CLINICAL TRIAL: NCT06730945
Title: A Multicenter, Randomized, Outcomes Assessor Blind, Parallel Controlled Trial to Evaluate the Effect of Oral Isosorbide Mononitrate Plus Amlodipine Antispasm Therapy on Outcomes of Radial Artery Grafts After Coronary Artery Bypass Grafting
Brief Title: Effect of Oral Isosorbide Mononitrate Plus Amlodipine Antispasm Therapy on Outcomes of Radial Artery Grafts After CABG
Acronym: ASRAB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Modify the trial design and construct a new larger trial.
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Professor and Director of Cardiovascular Surgery, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2025-XXX
Record Dates: First submitted 2024-12-07; First posted 2024-12-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Bypass Graft Surgery (CABG); Radial Artery Grafts; Graft Failure
Keywords: CABG; Radial artery grafts; Isosorbide Mononitrate; Amlodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isosorbide Mononitrate + Amlodipine (Experimental): Oral isosorbide mononitrate 40mg (if unable to tolerate, use 20mg) once daily + amlodipine 5mg (if unable to tolerate, use 2.5mg) once daily for 24 weeks after CABG
  Interventions: Drug: Oral isosorbide mononitrate 4+ amlodipine
- Blank control (No Intervention): no use of any nitrates or CCBs for 24 weeks after CABG. if there are indications of hypertension, use RAASi rather than CCB.

INTERVENTIONS:
Drug: Oral isosorbide mononitrate 4+ amlodipine — Oral isosorbide mononitrate 40mg (if unable to tolerate, 20mg) once daily + amlodipine 5mg (if unable to tolerate, 2.5mg) once daily for 24 weeks after CABG
  Arms: Isosorbide Mononitrate + Amlodipine

SUMMARY:
The goal of this clinical trial is to to evaluate the effect of oral isosorbide mononitrate plus amlodipine antispasm therapy on outcomes of radial artery grafts in patients underwent primary isolated CABG.

The main question it aims to answer is:

Whether the oral isosorbide mononitrate plus amlodipine antispasm therapy could reduce the failure outcome of radial artery grafts after CABG .

Researchers will compare isosorbide mononitrate plus amlodipine to none to see if isosorbide mononitrate plus amlodipine works.

Participants will

1. Take oral isosorbide mononitrate (20-40mg daily) plus amlodipine (2.5-5mg daily) therapy for 24 weeks after CABG.
2. Clinical follow-up at Week 1, 4, 12, and 24 after CABG.
3. Protocol-driven CCTA at Week 24 after CABG.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old，
* Any sex，
* Signed informed consent，
* Within 3 days after primary isolated CABG using RA graft

Exclusion Criteria:

1. Allergy to isosorbide mononitrate or amlodipine.
2. Hypotension (systolic BP <90 mmHg or diastolic BP <60 mmHg)
3. Acute myocardial infarction or cardiogenic shock
4. Contraindications for CCTA examination (eg., iodine allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The rate of RA graft failure at Week 24 | at Week 24
  A protocol-driven CCTA will be used to evaluate the RA graft outcome at Week 24 after CABG. Fitzgibbon Grade B/S/O is definned as Graft Failure.

SECONDARY OUTCOMES:
The time to first Major Adverse Cardiovascular Event (MACE) | within 24 weeks
  MACE is a composite of all-cause death, myocardial infarction（including peri-operative MI and silent MI), stroke and unplanned revascularization.
The proportion of participants with at least once symptomatic hypotension | within 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD, Principal Investigator — Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China; Mario FL Gaudino, MD, Principal Investigator — Weill Cornell Medicine NewYork Presbyterian Hospital, NY, US; Yunpeng Zhu, MD, Study Director — Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR